CLINICAL TRIAL: NCT06902090
Title: Safety, Tolerability and Pharmacokinetics of Meloxicam Nanocrystal Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yangtze River Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: YZJ-MLXK-PK-2207
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TR (Experimental)
  Interventions: Drug: Meloxicam Nanocrystal Injection(Yangtze River Pharmaceutical Group Co., Ltd.)
- Group RT (Active Comparator)
  Interventions: Drug: Meloxicam Nanocrystal Injection (ANJESO®)

INTERVENTIONS:
Drug: Meloxicam Nanocrystal Injection(Yangtze River Pharmaceutical Group Co., Ltd.) — IV, 30 mg
  Arms: Group TR
Drug: Meloxicam Nanocrystal Injection (ANJESO®) — IV, 30 mg
  Arms: Group RT

SUMMARY:
Primary Objective：To compare the pharmacokinetic profiles between meloxicam nanocrystal injection (strength: 1 mL: 30 mg, Yangtze River Pharmaceutical Group Co., Ltd.) and the originator meloxicam nanocrystal injection (trade name: ANJESO®, strength: 1 mL: 30 mg, Baudax Bio Inc.) in healthy volunteers.

Secondary Objective：To observe the safety and tolerability of meloxicam nanocrystal injection and ANJESO® in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to understand and willing to complete the study in strict compliance with the clinical protocol and sign the informed consent form.
2. Male or female subjects aged 18-45 years (inclusive), proper sex ratio.
3. Weight ≥ 50.0 kg for males, or ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (inclusive).
4. Subjects in good health, no respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system and other serious diseases or chronic disease history.
5. Subjects (including partners) have no donate sperm/eggs from 2 weeks before screening to 3 months after dosing, and voluntarily take appropriate contraceptive measures.

Exclusion Criteria:

1. Subjects who are known to be allergic to meloxicam, drug excipients or other NSAIDs, or have a history of two or more previous drug, food or pollen allergies, or a history of specific allergic diseases (such as asthma, urticaria, eczema, etc.).
2. Subjects who have special dietary requirements and cannot accept a unified diet.
3. Subjects who have poor peripheral venous access or cannot tolerate venous puncture or have a history of needle and blood fainting.
4. Subjects with clinically significant abnormalities as judged by the investigator based on results of physical examination, vital signs, 12-lead ECG, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function).
5. Those who are positive in any index screening of hepatitis B virus surface antigen, Treponema pallidum-specific antibody, human immunodeficiency virus antibody, or hepatitis C virus antibody.
6. Subjects with previous history (including existing) of gastrointestinal diseases (including gastrointestinal ulcers, gastrointestinal bleeding).
7. Subjects who have undergone major trauma surgery or have a history of trauma within 6 months before screening, or plan to undergo surgery during the study period.
8. Subjects with a history of drug abuse, drug use within 6 months before screening, or positive drug abuse screening.
9. Subjects who frequently consume alcohol within 3 months prior to screening, i.e., consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% spirits, alcohol or 150 mL of wine), or who cannot stop using any alcohol products during the study, or whose alcohol breath test result > 0.0 mg/100 mL.
10. Subjects who have donated blood or experienced massive blood loss (> 400 mL), received blood transfusions or used blood products within 3 months prior to screening.
11. Subjects who have consumed excessive tea, coffee and/or caffeine-containing beverages (more than 8 cups, 1 cup = 250 mL) daily during the 3 months before screening.
12. Subjects smoke an average of 5 or more cigarettes per day within 3 months prior to screening, or those who cannot stop using any tobacco products during the study.
13. Subjects who have participated in any clinical trial within 3 months prior to screening, or plan to participate in other clinical trials during the study.
14. Subjects who have received vaccination within 30 days prior to screening, or plan to receive vaccination during the study.
15. Subjects who have used any drugs that inhibit or induce hepatic metabolism of drugs (e.g., inducers - barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to screening.
16. Subjects who have taken any prescription drugs, over-the-counter drugs, health products, vitamins, and Chinese herbal medicines within 14 days before administration.
17. Subjects who have consumed special diets (including grapefruit, chocolate or xanthine-rich foods/beverages) within 48 h before administration.
18. Lactating women, or women who test positive for pregnancy.
19. Subjects with acute illness from screening period to pre-dose.
20. Subjects who should not be included in the investigator 's opinion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum drug plasma concentration) | up to 96 hours after drug administration
Tmax (Time to achieve Cmax) | up to 96 hours after drug administration
AUC0-t (Total area under the plasma drug concentration-time curve from time of administration to the time of the last quantifiable drug concentration) | up to 96 hours after drug administration
AUC0-∞ (Total area under the plasma drug concentration-time curve) | up to 96 hours after drug administration
T1/2z (Apparent terminal elimination half-life) | up to 96 hours after drug administration
λz (Apparent terminal elimination rate constant) | up to 96 hours after drug administration
AUC_%Extrap (The percentage of the portion estimated through extrapolation) | up to 96 hours after drug administration
Vz (Volume of distribution during the terminal phase) | up to 96 hours after drug administration
CLz (Clearance of the analyte in plasma) | up to 96 hours after drug administration
Occurence of adverse events | up to 5 days of each treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China